CLINICAL TRIAL: NCT03794817
Title: Immune Monitoring in Sensitized Patients at Risk of Rejection
Acronym: PRISM
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: PRISM
Record Dates: First submitted 2018-12-12; First posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Kidney Failure
Keywords: Kidney transplant recipient
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to test the effect of anti-rejection medications on your immune system

DETAILED DESCRIPTION:
Recipients of deceased or living donor transplants with calculated percent reactive antibody (cPRA) of 50% or greater at University of California, San Francisco (UCSF) will be enrolled in the trial. Samples for Kidney Solid Organ Response Test (kSORT) will be obtained pre-transplant (and immunosuppression) and post-transplant (see Table 1). Urine will be obtained at the same true intervals including pre-transplant in patients who still produce urine to correlate with graft rejection, inflammation and kSORT. A piece (minimum 1/3 core) of the protocol or for cause biopsy tissue will be saved in Ribonucleic acids (RNA) later for gene expression analysis as a correlate of graft inflammation with the biopsy, kSORT and urine. In addition, samples will be when patients are undergoing cause kidney biopsy, prior to treatment intensification and procedure. Patient's who are treated for rejection, will have additional samples obtained 2-4 weeks after treatment of rejection and at the time of any followup biopsy for monitoring resolution of biopsy confirmed acute rejection.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older able to consent
2. No history of HIV, hepatitis C and active hepatitis B infection
3. cPRA ≥ 50%

Exclusion Criteria:

1. Patients on Coumadin
2. Human Leukocyte antigen (HLA) identical donor recipient patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received a kidney transplant and will be taking immunosuppressive medications.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Immune monitoring in sensitized patients at risk of rejection | 2 years
  Pretransplant Kidney Solid Organ Response Test (kSORT) predictive value of rejection in the first 6 months after transplantation

SECONDARY OUTCOMES:
Kidney Solid Organ Response Test (kSORT) with pathological findings | 2 years
  Correlation of kSORT with pathological findings on kidney biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Vincenti, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No